CLINICAL TRIAL: NCT01519076
Title: A Feasibility Study: A Safety Evaluation of the Use of Magnetic-guided Iron Particles Administered to Patients Suffering Acute Ischemic Stroke and Treated With Tissue Plasminogen Activator (tPA)
Brief Title: A Safety Evaluation of the Use of Magnetic-guided Iron Particles
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Request
Sponsor: Pulse Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTI_CS001
Record Dates: First submitted 2012-01-18; First posted 2012-01-26 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Ischemic Stroke
Keywords: stroke
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Pulse Therapeutics (PTI) Magnetically-Enhanced Diffusion (MED) — The PTI MED System is a magnetic-controlled infusion system which uses external energy (magnetic energy) to drive an agent (tPA) to the desired target (blood clot).

SUMMARY:
This study is a prospective trial wherein each included subject will receive the experimental magnetically enhanced diffusion therapy. It will be conducted on a maximum of ten adult male or female patients who meet the inclusion and exclusion criteria and informed consent has been obtained. Subjects presenting in the emergency department with acute ischemic stroke and are eligible for tPA therapy may be considered for inclusion in the study.

DETAILED DESCRIPTION:
This study is a prospective trial wherein each included subject will receive the experimental magnetically enhanced diffusion therapy. It will be conducted on a maximum of ten adult male or female patients who meet the inclusion and exclusion criteria and informed consent has been obtained. Subjects presenting in the emergency department with acute ischemic stroke and are eligible for tPA therapy may be considered for inclusion in the study.

Subjects who meet the eligibility criteria will be treated with Magnetically Enhanced Diffusion (MED) concurrently with tPA infusion. Perfusion will be assessed using CTA/CTP at 2-4 hours upon completion of tPA infusion and using MRI at 24 hours upon completion of tPA infusion. Subjects are followed at 14 days, 30 days and 90 days post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between 18 and 80 years of age.
* Subject has moderate to large (NIHSS ≥ 10 and ≤24) ischemic stroke
* Subject has an intracranial arterial occlusion of the middle cerebral artery (MCA), anterior cerebral artery (ACA), internal carotid artery (ICA), posterior cerebral artery (PCA) or distal basilar artery confirmed by CT or MR angiography.
* Subject is eligible for initiation of intravenous tPA within three hours of stroke onset, where time of stroke onset is defined as the last time the patient was witnessed to be at baseline.

Exclusion Criteria:

* Subject has known sensitivity to iron or PEG products.
* Subject has recently (within 30 days) received iron replacement therapy.
* Subject has known or suspect liver function abnormality.
* Subject has known or suspect severe renal impairment.
* Subject has a high-density lesion on baseline CT scan consistent with hemorrhage of any degree.
* Subject has a significant mass on baseline CT consistent with midline shift.
* Subject has a large (greater than one-third of the middle cerebral artery) regions of clear hypodensity on the baseline CT scan.
* Subject has evidence of intraparenchymal tumor on baseline CT scan.
* Subject experiences a seizure at the onset of stroke.
* Subject has known hemosiderosis or hemochromatosis.
* Subject has an implantable cardioverter defibrillator, pacemaker, neurostimulator or other device incompatible with MRI.
* Subject has a history of stroke within the last three months.
* Subject has a previous or existing intracranial hemorrhage, neoplasm, subarachnoid hemorrhage or arteriovenous malformation.
* Subject has experienced any active or recent (within 30 days) hemorrhage.
* Subject has systolic blood pressure > 185 mmHg or diastolic > 110 mmHg.
* Subject has presumed septic embolus or suspicion of bacterial endocarditis.
* Subject has presumed pericarditis including pericarditis after acute myocardial infarction.
* Subject is suspected to have an aortic dissection.
* Subject has recently (within 30 days) undergone surgery or biopsy of a parenchymal organ.
* Subject has recently (within 30 days) experienced trauma with internal injuries or ulcerative wounds.
* Subject has recently (within 90 days) experienced severe head trauma with loss of consciousness.
* Subject has known hereditary or acquired hemorrhage diathesis, coagulation factor deficiency, or oral anticoagulant therapy with INR > 1.7 or institutionally equivalent prothrombin time.
* Subject has a glucose level of < 50 mg/dl or >400 mg/dl, or a platelet count less than 100,000, or an Hct level less than 25.
* Subject has taken dabigatran within the last 48 hours or any new anticoagulant which cannot be monitored by traditional.
* Subject requires hemodialysis or peritoneal dialysis, or has a contraindication to angiogram.
* Subject has prolonged partial thromboplastin time (PTT) (in the case where heparin or a direct thrombin inhibitor has been administered within 48 hours).
* Subject has had a recent (within 7 days) lumbar puncture or arterial puncture at a non-compressible site.
* Subject has a pre-existing neurological or psychiatric disease that would confound evaluations.
* Subject is pregnant, nursing or intends to become pregnant during the trial period.
* Subject is currently enrolled in other potentially confounding research.
* Subject has any condition that, at the discretion of the investigator, would preclude participation in the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-06; Primary Completion 2014-01 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Safety: incidence and evaluation of any adverse effects associated with the investigational procedure compared with historical controls treated with tPA alone. | 90 days
  The primary measures of safety will be mortality at 3 months and symptomatic ICH within the first 24 hours post-treatment. All intracerebral hemorrhages (ICH) will be classified radiographically using the ECASS criteria. The proportion of subjects with Type II parenchymal intracerebral hematomas within the first 24 hours post-treatment and the incidence of any asymptomatic hemorrhage within the first 24 hours will also be compared.

SECONDARY OUTCOMES:
Brain Recanalization and perfusion | 24 hours
  The degree of recanalization (partial and complete) and reperfusion will be assessed at 2-4 hours post-treatment using CT angiography, and at 24 +/- 6 hours post-treatment using MRI. TIMI Grade Flow of 2 or 3 will be considered "responsive to treatment".

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Bladin, MD, Principal Investigator — Eastern Health Services Box Hill Hospital
Locations (2):
- Australia (2):
  - Hunter New England, New Lambton, New South Wales
  - Eastern Health Services Box Hill Hospital, Box Hill, Victoria